# Montefiore Medical Center Albert Einstein College of Medicine of Yeshiva University Individual's Informed Consent to Participate as a Subject in Clinical Research

You are being asked to join this research study.

The title of the study is: Prospective tissue collection in breast cancer patients receiving preoperative systemic therapy.

The study is being done under the supervision of:

Principal Investigator (Researcher Study Doctor): Jesus Anampa-Mesias, MD

Office Address: 1695 Eastchester Road 2<sup>nd</sup> Floor, Bronx, NY 10461

Telephone #: 718-405-8404 IRB Protocol #: 13-02-079

### DO I HAVE TO TAKE PART IN THIS RESEARCH STUDY?

- Your participation is voluntary. This means that you decide whether you want to join the study after speaking with the researcher, or other members of the research team.
- If you decide to take part, you will be asked to sign this consent form. Your signature means that you agree to be a subject in this research.
- After reading this form and discussing what it says, you should ask all the questions you want to ask. You should take as much time as you need to decide.
- If you do not understand some of the terms used in this form, ask the person who is discussing the study with you to give any additional information that may make this easier to understand.
- You do not have to consent to participate in the study immediately, or ever. Take time to decide whether you wish to join. You may take home a copy of this consent form to think about it or discuss the information with family or friends before you decide.
- If you decide not to participate the care providers at this facility will give you all the standard care that is appropriate for you.
- You will be given a copy of this form whether you agree to participate in this study. Do
  not sign the form unless you have had all your questions answered and understand
  exactly what is involved.
- If you decide to take part, you are still free to withdraw at any time without giving a reason. This will not affect your care and you will continue to be treated at this facility.
- If you decide to withdraw after receiving the study drug, you should talk with the research study doctor to see how best to complete the withdrawal process.
- The form discusses:

WHAT THE RESEARCHERS WILL LEARN FROM THE RESEARCH WHAT WILL HAPPEN TO YOU DURING THE RESEARCH WHAT RISKS AND/OR DISCOMFORTS YOU MIGHT EXPECT/EXPERIENCE AS A RESEARCH SUBJECT

IF YOU CAN EXPECT ANY BENEFITS AND ARE THERE ANY ALTERNATIVES TO THIS RESEARCH FOR YOUR CONDITION.

### WHY HAVE I BEEN ASKED TO TAKE PART IN THIS RESEARCH STUDY?

• You are being asked to take part in this study because you have breast cancer\_that has a high chance of having spread to other organs if treated by surgery alone.

### WHY IS THIS RESEARCH STUDY BEING DONE?

This study involves blood and/or tissue collection during treatment with **standard** chemotherapy for the treatment of breast cancer.

The purpose of this study is to obtain blood and/or tumor samples before treatment, 2-3 weeks after treatment begins and before surgery to find tests that may lead to a better understanding of how the chemotherapy is working and might predict which patients will or will not respond to chemotherapy. This may help to develop better treatments in the future.

### HOW MANY PEOPLE WILL TAKE PART IN THE RESEARCH STUDY?

With reopening of the study, a total of 92 patients will take part in this study, all at Montefiore Medical Center.

### WHAT WILL HAPPEN IF I TAKE PART IN THIS RESEARCH STUDY?

You will be treated with the <u>same standard chemotherapy combinations used most commonly for patients who are not participating in a research study</u>. The combination of chemotherapies will depend on the type of breast cancer that you have.

If the breast cancer is HER2 negative (about 75% all cancers), then you will be treated with paclitaxel (+/- carboplatin) given weekly for 12 weeks followed by doxorubicin and cyclophosphamide given every 2 -3 weeks for 4 treatments, or you will be treated with the same drugs in the reverse sequence if your doctor feels that is a better tolerated sequence in your case. Both sequences are considered standard ways to administer this treatment. Other standard of care chemotherapy regimens can be used as per your physician decision such as docetaxel plus cyclophosphamide, or docetaxel plus carboplatin. Pembrolizumab can be used in patients who have HER negative/ER negative disease. If your tumor is estrogen-receptor (ER) positive and your doctor feels you are a good candidate for hormonal therapy, you will have a 4-6 month or longer course of hormonal therapy prior to surgery.

You will receive tests and examinations that are routinely used for the treatment of breast cancer.

The study procedures are summarized below:

- **Before treatment:** Blood specimens (3-5 tubes, about 3-5 tablespoons). Fine needle aspiration (FNA) of the breast tumor (5 passes using a thin needle) is recommended, but is <u>optional</u>. A sample from the biopsy that was done to diagnose breast cancer will be collected.
- **After 2-3 weeks on study:** Blood specimens (3-5 tubes, about 3-5 tablespoons). Fine needle aspiration (FNA) of the breast tumor (5 passes using a thin needle) is

recommended but is optional.

• At the time of Surgery: Blood specimens (3-5 tubes, about 3-5 tablespoons). A sample of breast tumor removed at time of surgery will be collected.

### WILL THIS STUDY INVOLVE GENETIC RESEARCH and/or TESTING?

Genetic means having to do with information that is passed on in families from parents to their children through genes.

No, this study will not involve genetic research and/ or testing.

In the future, before the extract from your tissue or blood samples can be used for research, the people doing the research must get a specific approval from the Institutional Review Board (IRB) of Montefiore/Einstein. The IRB is a committee made up of doctors, researchers and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at Montefiore/Einstein, including research involving your tissue and blood samples from this bank must first be approved by the IRB. Portions of the extracts from the tumor specimens and blood samples may be shared with investigators outside Montefiore/Einstein in order to perform studies on the tissue that are not readily available at this institution.

**Treatment** (explained in detail in the next several paragraphs):

You will not need to be hospitalized to take part in this study.

The standard of care treatment, <u>not related to this study</u>, will include excision of your tumor that may require hospitalization and standard chemotherapy, Your doctor may choose one of the following standard treatment options that he/she thinks is the best option for you based on its effectiveness and side effect profile:

### **Stratum I (HER negative, chemotherapy indicated)**

Patients in Stratum I can be treated with the following regimens:

### If hormone positive:

- Paclitaxel weekly x12 consecutive weeks followed by AC every 2 weeks for 4 cycles, OR
- Docetaxel plus cyclophosphamide IV every 3 weeks for 4-6 cycles, OR

### If hormone negative:

- Paclitaxel weekly x12 weeks (+/- carboplatin) followed by AC every 2-3 weeks x4 cycles, OR
- Docetaxel plus cyclophosphamide IV every 3 weeks for 4-6 cycles, OR
- Docetaxel plus carboplatin IV every 3 weeks for 4-6 cycles.
- If there is no contraindication to immunotherapy, ER- patients will receive pembrolizumab every 3 weeks for 6-8 doses along with neoadjuvant chemotherapy.

### Stratum II (Hormone positive, Her2 negative, Endocrine therapy indicated)

Patients in Stratum II can be treated with the following regimens:

- Anastrozole 1 mg po daily for 4-6 months.
- Letrozole 2.5 mg po daily for 4-6 months.
- Exemestane 25 mg po daily for 4-6 months.
- Tamoxifen 20 mg po daily for 4-6 months.

#### When I am finished taking the standard chemotherapy

- You will undergo breast surgery. The surgery may include a mastectomy or lumpectomy, whichever procedure your research study doctor feels is the best procedure to remove the breast tumor. Most patients with locally advanced breast cancer require mastectomy in order to assure that all the tumor cells have been removed. The surgery will usually also include removal of the axillary lymph nodes (lymph nodes in the arm pit). Your research study doctor will ask you to sign a separate hospital consent form for the surgery. Potential complications from the surgery include pain, bleeding, and infection.
- Your surgical and blood specimen will be collected for mandatory research studies.
- You will follow up in 3-4 weeks with the study doctor.
- If you developed side effects, shown either by physical exam or laboratory abnormalities, your doctor will continue to follow you until resolution of these issues.
- Standard post-operative care will continue. After completing the protocol-specified therapy indicated above, your research study doctor may advise additional treatment that is part of routine standard care. These possible treatments include radiation therapy, hormonal therapy, and continued trastuzumab therapy. These are considered standard treatments and are not part of this research study. If radiation therapy is given, it typically begins within about 4 weeks of completion of chemotherapy. You will be evaluated by a radiation oncologist who will discuss the potential benefits and

risks of radiation, and who will prescribe and monitor the radiation. It is usually given as a single dose to the breast, chest wall, and nearby lymph nodes five days per week for 6 weeks.

- If your tumor is estrogen-receptor (ER) positive, your research study doctor will also recommend hormonal therapy (e.g., tamoxifen or an aromatase inhibitor [such as anastrozole, letrozole, or exemestane]) for a period of at least 5 years, or possibly longer.
- If you received pembrolizumab prior to surgery, you will be treated with the same drug for up to 27 weeks after surgery.
- If your disease still remains after surgery, you will be treated with capecitabine.
- If you have germline BRACA1/2 mutation and HER2 negative tumors who meet standard of care guidelines, you will be given PARP inhibitors after surgery.
- If you have high-risk HR+/HER2 breast cancer which meets standard of care guideline, you will be given abemaciclib.

### **Study Plan**

Another way to find out what will happen to you during the study is to read the chart below. Start reading at the top and read down the list, following the lines and arrows.





### WHAT ELSE DO I HAVE TO DO?

- You must tell the research study doctor about any past and present diseases or allergies
  you are aware of and about all medications you are taking including over-the-counter
  remedies and nutritional supplements or herbs.
- If you do not feel well at any time, call your doctor or the research study doctor immediately.
- Drugs may cause a reaction that, if not treated promptly, could be life-threatening. It is important that you report all symptoms, reactions and other complaints to the research study doctor.
- If you think you have become pregnant, contact your research study doctor immediately.
- If any other doctor recommends that you take any medicine, please inform him/her that you are taking part in a research study. You should give the other doctor the research study doctor's name and phone number.
- You may carry out all your normal daily activities that are suitable to you.

### **HOW LONG WILL I BE IN THE STUDY?**

You will be asked to take <u>standard pre-operative chemotherapy</u> treatment for 18-24 weeks. Treatment may be stopped if:

- your tumor progresses (grows) despite the treatment.
- you develop severe side effects.
- scientific developments occur that indicate the treatment is not in your best interest or
- you elect to withdraw from the research protocol for any reason.

After you are finished taking pre-operative treatment, you will undergo surgery. Following the surgery, the study doctor will ask you to visit the office for follow-up exams every 6 months for the first 5 years and yearly for the next 5 years. We would like to keep track of your medical condition for the rest of your life. We would like to do this by calling you on the telephone once a year to see how you are doing. Keeping in touch with you and checking on your condition every year helps us look at the long-term effects of the study.

### WHAT ARE THE POSSIBLE SIDE EFFECTS, DISCOMFORTS, RISKS OR INCONVENIENCES I CAN EXPECT FROM BEING IN THIS RESEARCH STUDY?

**<u>Blood Drawing</u>**: This may cause temporary bruising and pain at the puncture site. There is also the possibility you may experience bleeding into the tissue around where the blood was drawn, and an infection may occur.

**Fine Needle Aspiration (FNA):** Having an FNA biopsy performed may cause mild pain (very common), bruising (occasional), bleeding (rare), redness (rare), swelling (rare), and/or infection (extremely rare) at the site of the biopsies. Mild pain is usually controlled with over-the-counter pain relievers. Most side-effects go away within a few days.

If infection occurs with either of the procedures, it will be treated accordingly with the standard of care antibiotics.

Everyone taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen. You should talk to your study doctor about any side effects that you have while taking part in the study. Your health care team may give you medicines to help lessen side effects. Many side effects go away soon after you stop taking the standard treatment. Death as result of FNA or blood draw is very rare.

### PREGNANCY AND IMPREGNATION DURING THIS STUDY

- The drug(s) used to treat breast cancer are not part of the study. You should discuss with your medical oncologist about the implications of pregnancy in the treatment of breast cancer.
- For more information about risks and side effects, ask your research study doctor.

### ARE THERE LIKELY TO BE ANY BENEFITS TO TAKING PART IN THIS RESEARCH STUDY?

If you take part in this study, there will be no medical benefit to you. We hope the information learned from this study will benefit other breast cancer patients in the future.

### WHAT OTHER CHOICES DO I HAVE IF I DO NOT TAKE PART IN THIS RESEARCH STUDY?

Before agreeing to join the study and before signing this consent form your personal doctor should have discussed with you what, and if, standard treatments are available and/or other research protocols. Your other choices may include:

- Getting similar treatment or care for your cancer without being in a research study.
- You may choose not take part in this study and take part in another study.

Talk to your research study doctor about your choices before you decide if you will take part in this study.

#### WILL I BE PAID FOR BEING IN THE STUDY?

You will not be paid for taking part in this research study.

#### WHO MAY SEE MY RECORDS?

- The research records will be kept private, and your name will not be used in any written or verbal reports.
- Your research records and medical records may be inspected by members of the research team and designated employees of Montefiore Medical Center.

- As this research involves a drug, the U.S. Food and Drug Administration (FDA), the agency for regulating the drugs, may inspect your research records and medical records.
- The research study doctor and research staff will review your medical records and will keep the information private.
- All laboratory specimens, reports, and other records will be identified only by a number known only to the research study doctor. The research records will be kept in a secured manner and computer records will be password protected.
- The people who reviewed this research study as members of the Institutional Review Board of The Albert Einstein College of Medicine may also review your research and medical records.
- The Office for Human Research Protections (OHRP) may also review your research study records.
- All of these groups have been requested to keep your name private.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This Web site will not include information that can identify you. At most, the Web site will include a summary of study results. You can search this Web site at any time.

#### WILL THERE BE ANY COSTS TO ME?

You and/or your health plan/ insurance company will need to pay for some or all of the costs of treating your cancer in this study. Some health plans will not pay these costs for people taking part in studies. Check with your health plan or insurance company to find out what they will pay for. Taking part in this study would not cost your insurance company more than the cost of getting regular cancer treatment. All treatment agents are commercially available and all tests (with the exception of the tumor biopsy and research blood specimens) are considered standard of care for your condition.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

### WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THIS RESEARCH STUDY?

If there is a physical injury as a result of this research, only immediate, essential, short-term medical treatment as determined by the participating hospital, will be available for the injury without charge to you personally.

- No monetary compensation will be offered.
- You are not waiving any of your legal rights by signing this informed consent document.
- If additional treatment is required as a result of a physical injury related to the research, necessary medical treatment will be provided to you and billed to your insurance company or to you as part of your medical expenses.

Immediately report any discomforts, problems or injuries you experience during the course of your participation in the study to Dr. Jesus Anampa at 718-405-8404.

### WHO CAN ANSWER MY QUESTIONS ABOUT THE STUDY?

Researcher's Name: Dr. Jesus Anampa

Office Address: Montefiore Einstein Cancer Center1695 Eastchester

Rd, Bronx, NY 10461

Office Phone: 718-405-8404

- If any questions arise related to this research project, or you believe you have any injury related to this study, you can call the researcher above.
- You may also call Anastasia Abdul -Wahab at 718-405-8505.
- If you have questions regarding your rights as a research subject, you may also call the Administrator of The Albert Einstein College of Medicine Institutional Review Board (IRB) at (718) 798-0406, Monday through Friday between 9 AM and 5 PM.

### WHERE CAN I GET MORE INFORMATION?

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You will get a copy of this form. If you want more information about this study, ask your study doctor.

### WILL ANY OF THE SAMPLES (BLOOD, TISSUE, DNA) TAKEN FROM ME BE USED FOR FUTURE RESEARCH STUDIES?

In addition to the research you are consenting to under this research study, Dr. Jesus Anampa or other researchers at this or other institutions may wish to study the samples in future research, which unlikely may include genetic analysis. These samples, taken from your body, would NOT be linked back to you. No one will know your name or protected health information.

At this time, the researcher does not know what the future studies will be. Your specimens may also be submitted to a tissue/cell/DNA bank. The specimens may be kept for a long time and may be more than 50 years.

In some research using human blood or tissue, the specimens and their parts may enable researchers to develop medical tests or treatments that have commercial value. You will not receive any money that may result from any such commercial tests or treatments.

Your specimens may be used for future research, even though the purpose of the future research is not known at this time.

## PARTICIPANT: PLEASE INDICATE YOUR CHOICE BY INITIALING ONE (1) OF THE FOLLOWING OPTIONS

| I consent to have my specimens used for future research studies. | V CINRBIEXPIRM HON, BAYFE; 10/ |
|---|---|
| I consent to have my specimens used for future research studies | only for the study of |
| I do NOT consent to have my specimens used for future research will be destroyed at the end of the study.) | studies. (The specimens |

## <u>CAN I BE ASKED TO STOP PARTICIPATING IN THIS STUDY BEFORE THE</u> STUDY IS FINISHED?

Sometimes the company sponsoring the research may stop your part in the study for the following reasons:

- You fail to follow instructions given to you by the research study doctor.
- New information about important medical risks and benefits become available.
- If you are a female and become pregnant while on the study, you will be taken off of protocol treatment.

### WHAT IF NEW INFORMATION BECOMES AVAILABLE?

- If the research study doctor obtains new information that might lead you to change your mind about continuing in this study, the research study doctor will tell you about it.
- If you decide to withdraw, the research study doctor and your personal doctor will make arrangements for your care to continue.

### MAY I STOP THE STUDY AT ANY TIME?

- Your participation in this study is voluntary, and you may withdraw from the study at any time without giving a reason.
- It is important to tell the study doctor if you are thinking about stopping so any risks from the treatment or biopsies can be evaluated by your doctor.
- If you agree to participate and withdraw at a later time, some of your information may have already been entered into the study and that will not be removed.
- In addition, you may be asked to return to the research study doctor again for any final tests in order to close the record and tests or monitoring that are necessary for your health as a result of your participation. These results may be recorded.
- Your treatment by doctors and staff at the institution(s) involved in this study, now and in the future, will not be affected in any way if you agree to participate and withdraw later.

### WHAT ARE MY RIGHTS IF I TAKE PART IN THIS RESEARCH STUDY?

- Your participation in this study is voluntary.
- You do not waive any of your legal rights by participating in this research study.
- Your treatment by doctors and staff at the institution(s) involved in this study, now and in the future, will not be affected in any way if you refuse to participate or if you enter the study and withdraw later.

### **Informed Consent Signature Page**

The following is a list of items that have been discussed with you about this research study. If you have any questions about any of these items, please ask the person who is discussing the study with you for more information before agreeing to participate.

- What the study is about.
- What I must do when I am in the study.
- The possible risks and benefits to me.
- Who to contact if I have questions or if there is a research related injury.
- Any costs and payments.
- I can discontinue participating in the study at any time without penalty.
- Other choices.
- My name will not appear on interview or other data collection forms.
- All written and published information will be reported as group data with no reference to my name.
- If there is a schedule explaining how the study medicines are to be taken, I will be given the time schedule.
- I have been given the name of the researcher and others to contact.
- I have the right to ask any questions.

| Optional Procedure | | Patient<br>Initials | Date |
|---|---|---|---|
| I consent to have a Fine Needle Aspiration of the tumor for research before therapy (initial and date if yes) | | | |
| • I consent to have a Fine Needle Aspiration of the tumor for research after 2-3 weeks after therapy begins (initial and date if yes) | | | |
| Printed Name of Participant | Signature of Participant | | Time |
| Printed Name of Person Conducting the Informed Consent Process | Signature of Person Conducting the Informed Consent Process | Date | Time |